CLINICAL TRIAL: NCT03514498
Title: Cognitive, Behavioural and Metabolic Effects of Anesthesia in Patients With Autism Spectrum Disorder: a Pilot Study
Brief Title: Autism & Anesthetic Exposure Study
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Mark Crawford, Anesthesiologist-in-Chief, The Hospital for Sick Children
Other Study IDs: 1000057105
Record Dates: First submitted 2018-03-29; First posted 2018-05-02 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Autism Spectrum Disorder
Keywords: anesthesia
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell lines will be established from blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder: Children aged 4-12 years with a clinical diagnosis of mild-to-moderate Autism Spectrum Disorder undergoing dental surgery
  Interventions: Procedure: Dental surgery
- Typically Developed Controls: Children with no neurodevelopmental delays matched to Autism Spectrum Disorder participants according to age (within 6 months), gender, and ASA physical status level, scheduled to undergo dental surgery
  Interventions: Procedure: Dental surgery

INTERVENTIONS:
Procedure: Dental surgery — All types of dental surgery

SUMMARY:
As anesthesia is often needed for childhood surgery and procedures, researchers have examined the potential effects of anesthesia on neurodevelopment. There are few studies that have examined the effect of anesthesia on neurodevelopment in children with confirmed diagnoses of ASD, and the results of these studies are mixed. Children with neurodevelopmental disorders can have age-dependent variations in brain anatomy, function, and connectivity, which may alter their sensitivity to the potential neurotoxic effects of anesthetic and sedative drugs. Given the potential adverse neurodevelopmental effects of anesthesia on typically developing children, it is important to examine if anesthesia exposure can worsen the clinical course of ASD.

DETAILED DESCRIPTION:
We hypothesize that children with a confirmed diagnosis of ASD will regress developmentally following general anesthesia for dental surgery in comparison to children without ASD (controls) undergoing dental surgery. In this pilot study, we will investigate this hypothesis through the following objectives:

1. to determine in a clinical study if anesthesia induces post-operative persistent adverse changes children with ASD as compared with typically developing controls;
2. to determine the potential mechanism for the adverse effects of anesthetics on patients with ASD compared to healthy controls, peripheral blood mononuclear cells will be isolated from blood samples (PBMCs), before genomic DNA isolation for mitochondrial content analysis.

ELIGIBILITY:
Inclusion Criteria For Autism Spectrum Disorder Group:

* child is undergoing dental surgery
* child is aged 4 to 12 years
* child has mild-to-moderate diagnosis of autism spectrum disorder
* child has an American Society of Anesthesiologists (ASA) Physical Status level I or II

Exclusion Criteria for Autism Spectrum Disorder Group:

- child does not use words or phrases to communicate

Inclusion Criteria for Typically Developed Controls Group:

* child is undergoing dental surgery
* child is matched to an autism spectrum disorder participant according to age, gender, and ASA level

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children undergoing dental surgery at The Hospital for Sick Children
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Current language and behaviour skills | up to 3 months before surgery
  measured using the Autism Diagnostic Interview - Revised
Regression in language and behaviour skills | up to 12 weeks following anesthetic exposure
  measured using the Autism Diagnostic Interview - Revised

SECONDARY OUTCOMES:
Metabolic make-up | immediately prior to anesthetic exposure
  measured using quantitative polymerase chain reactions
Metabolic changes | within 1-2 hours following anesthetic exposure
  measured using quantitative polymerase chain reactions
Current non-specific behaviour skills | up to 3 months before surgery
  measured using the Abberant Behaviour Checklist
Regression in non-specific behaviour skills | up to 12 weeks following anesthetic exposure
  measured using the Abberant Behaviour Checklist
Current sleep habits | up to 3 months before surgery
  measured using the Children's Sleep Habits Questionnaire
Regression in sleep habits | up to 12 weeks following anesthetic exposure
  measured using the Children's Sleep Habits Questionnaire
Current social communication skills | up to 3 months before surgery
  measured using the Social Communication Questionnaire
Regression in social communication skills | up to 12 weeks following anesthetic exposure
  measured using the Social Communication Questionnaire
Current social responsiveness skills | up to 3 months before surgery
  measured using the Social Responsiveness Scale
Regression in social responsiveness skills | up to 12 weeks following anesthetic exposure
  measured using the Social Responsiveness Scale
Posthospitalization Behaviours | 3 days following anesthetic exposure
  measured using the Posthospitalization Behaviour Questionnaire
Changes in posthospitalization behaviours | up to 12 weeks following anesthetic exposure
  measured using semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Mark Crawford, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No